CLINICAL TRIAL: NCT05703633
Title: Single Center, First-In-Man, Proof-of-Concept Study: Transplantation of Uncontrolled DCD Kidneys REconditioned by a Novel Ex-VIVo Perfusion MEthod - The REVIVEME Trial
Brief Title: Transplantation of Uncontrolled DCD Kidneys REconditioned by a Novel Ex-VIVo Perfusion MEthod
Acronym: REVIVEME
Status: Unknown | Phase: Phase 1 / Phase 2 | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Sahlgrenska University Hospital (Other)
Responsible Party: Principal Investigator, Michael Olausson, Professor, Sahlgrenska University Hospital
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: GOT.2023.1
Record Dates: First submitted 2023-01-19; First posted 2023-01-30 (Actual); Last update posted 2023-01-31 (Actual); Status verified 2023-01

CONDITIONS: End-Stage Kidney Disease
Keywords: Kidney Transplantation; uDCD
MeSH Terms: conditions — Kidney Failure, Chronic

STUDY DESIGN:
Intervention Model Description: Single center, open label, proof-of-concept study, Phase 1-2a
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- uDCD arm (Experimental): Patients enroled in the study will receive a kidney from a uDCD donor, after the kidney has been subjected to a reconditioning procedure, preventing ischemia/reperfusion-injury, confirming large animal data using the same protocol.
  Interventions: Other: uDCD treatment

INTERVENTIONS:
Other: uDCD treatment — Thrombolytic treatment/prevention ex-vivo to kidneys procured from patients after circulatory arrest

SUMMARY:
Eight patient will be transplanted with kidneys from donors dying after uncontrolled circulatory arrest (uDCD), with prolonged warm ischemia (up to 4,5 hours), preserved by a new method based on removal of fibrinogen/fibrin in the capillary systems, leading to an effective oxygenation of the tissue using an ex-vivo hospital manufactured perfusion device, minimizing the risk for ischemia-reperfusion injury (I/R-I) after kidney transplantation.Each patient will be studied for three months, with long-term follow-up data collected at 6 and 12 months

DETAILED DESCRIPTION:
In a large animal model the investigators have shown that kidneys from uDCD donors, subjected to 4½ hours of warm ischemia time (WIT) can be safely reconditioned to normal function, without the use of advanced cardiopulmonary resuscitation (aCPR), extracorporeal circulation, or use of anticoagulants given to the donor. Furthermore, kidneys from uDCD, treated according to the new method, can safely be transplanted into pigs, having normal renal function (measured with creatinine and iohexol-clearance) at the three-month follow-up. Toxicity studies in pigs, conclude that minimal amounts of drugs are transferred at the transplantation, most of the components being reduced during the ex-vivo process, showing levels transferred to the recipient being very low. The renal histology was close to normal in biopsies taken from the kidneys surviving three months, without signs of fibrosis or glomerulosclerosis. Our research is supported by data from other labs. In short - our new method means that the investigators prevent the I/R-I caused by obstruction of the arterial flow, with hypoxia as result. Normally, at reperfusion, fibrin in abundance will result in clot formation when activated platelets and red blood cells (RBCs) arrive. Consequently, kidneys will tolerate a substantially longer WIT than if the capillaries would have been occluded with hypoxia as result. Based on our large animal data, the investigators have strong reasons to believe that the proposed new method significantly will reduce the frequency of delayed graft function (DGF), increase the quality of the renal grafts, and increase the donor pool for successful kidney transplantations.

The present study protocol describes a first-in-human trial, in which uDCD-kidneys are reconditioned and preserved using this new perfusion method and then transplanted to patients on the waiting list for diseased donors. The purpose of the present clinical proof-of-concept (PoC) trial is to show that a novel method for preservation of donated kidneys with prolonged warm ischemia time, developed in pigs, can be safely transferred to transplantations of uDCD-kidneys in humans.

Injection time of Solution A is defined as the start of the reconditioning phase. Solution A is injected into the renal arteries of the explanted kidneys after closing the renal veins with a vascular clamp. A clamp is placed on the arteries after injection of Solution A. After 30 to 210 min, a second dose of Solution A is given, followed by Solution B 15 min later, injected into the renal arteries. During the next 15 -30 minutes, vascular adapters for the aorta patches/arteries and nipples for the ureters are mounted. The kidneys are moved to the organ chamber in a hospital manufactured medical technical product (MTP) and connected to the perfusion circuit. The oxygenated perfusion is started at 24 °C at a pressure of 30 mmHg. The pressure is gradually increased with 5 mmHg every minutes up to a maximum of 80 mmHg, to allow for the capillaries to be cleared of fibrin clots, after which temperature is decreased to 15 °C and the pressure to 20mmHg. After three hours, washed RBCs (with low platelet counts) are added, temperature is raised to 25 mmHg and temperature to 28-32 °C. Oxygenated perfusion is continued, with the perfusate passing through adsorbers. Vascular resistance and flow are monitored for during the whole medical device perfusion process. After final evaluation and assessment of the kidneys by the user, temperature is decreased to 15 °C and pressure to 20 mmHg, with perfusion continuing until kidney is disconnected and retrieved from the organ chamber and assessed for viability for transplantation by the user prior to being transplanted.

ELIGIBILITY:
Inclusion Criteria:

* Both sexes
* Age 18 - 65
* First-time transplant
* ABO blood-group identical
* Living within 4 hours from transplant site
* Written consent

Exclusion Criteria:

* Human Leukocyte Antigen (HLA) antibodies and/or preformed donor specific antibodies (DSA)
* Total ischemia time of > 16 hours
* Multi organ transplant recipients or previously transplanted
* ABO-incompatible or positive complement-dependent crossmatch (CDC X-match)
* Contraindicating medical condition
* Contraindicating malignancy
* Recent drug abuse
* Non-adherent or difficulties understanding the protocol
* Known risk factors for technical surgical complications (i.e. serious arteriosclerosis and or obesity)

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 8 (Estimated)
Dates: Start 2023-08-21 (Estimated); Primary Completion 2024-08-31 (Estimated); Study Completion 2024-12-31 (Estimated)

PRIMARY OUTCOMES:
Safety - Serious Adverse Events | Three months post transplantation
  Occurrence of serious adverse events, Clavien-Dindo IV-V grade complications, including primary none function

CONTACTS AND LOCATIONS:
Overall Officials: Niclas Kvarnström, MD, PhD, Study Chair — Västra Götalandsregionen - SU - Sahlgrenska

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Olausson M, Antony D, Travnikova G, Johansson M, Nayakawde NB, Banerjee D, Softeland JM, Premaratne GU. Novel Ex-Vivo Thrombolytic Reconditioning of Kidneys Retrieved 4 to 5 Hours After Circulatory Death. Transplantation. 2022 Aug 1;106(8):1577-1588. doi: 10.1097/TP.0000000000004037. Epub 2022 Jul 22. PMID 34974455
- [Background] Olausson M, Antony D, Johansson M, Travnikova G, Nayakawde NB, Banerjee D, Mackay Softeland J, Ognissanti D, Andresen Bergstrom M, Hammarsten O, Premaratne GU. Long-term Transplant Function After Thrombolytic Treatment Ex Vivo of Donated Kidneys Retrieved 4 to 5 H After Circulatory Death. Transplantation. 2022 Dec 1;106(12):2348-2359. doi: 10.1097/TP.0000000000004235. Epub 2022 Nov 22. PMID 35831928